CLINICAL TRIAL: NCT05580315
Title: EPOS Discoid Meniscus (DiMe) Project: a Prospective Multicentric Cohort Protocol
Brief Title: EPOS Discoid Meniscus (DiMe) Project
Acronym: DiMe
Status: Recruiting | Type: Observational
Sponsor: University of Milano Bicocca (Other)
Responsible Party: Sponsor
Other Study IDs: DiMe
Record Dates: First submitted 2022-10-04; First posted 2022-10-14 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Discoid Meniscus of Knee
Keywords: discoid meniscus; knee; pediatric; sport medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The aims of this Discoid Meniscus (DiMe) project are to analyze DM tears characteristics in the pediatric European population to describe current treatment options in symptomatic DM, and to evaluate clinical outcomes. To reach these objectives, a prospective database including symptomatic DM and variables associated with DM characteristics, type of tears, treatment, imaging, and clinical follow-up will be implemented. Data collection platform will provide future studies to understand the best treatment option for skeletally immature patient with symptomatic DM according to their history and lesion characteristics.

DETAILED DESCRIPTION:
This is a multicentric international prospective cohort study. All eligible consecutive patients will be identified prospectively by the local participating clinical teams according to Inclusion/Exclusion Criteria. Prospective data entry is mandatory.

Data collection will be conducted in three phases:

* Phase 1 will register patients to the study, document symptomatic DM, collect the details of patient demographics, sport characteristics, PROMS, imaging classification and consent of the patient's legal representatives. Once the patient has reached the age of majority, the date of his/her own consent will be recorded.
* Phase 2 will register surgical treatment and arthroscopic video and photographs collected during surgery, collect intraoperative DM instability, arthroscopic classification, and surgical details. Post-operative complication will also be collected.
* Phase 3 will collect short-, medium- and long-term outcome data. Short follow-up data collection will plan at 1 month follow-up then 3 and 6-months follow-up. Then annual data collection will be performed.

The foreseen timeframe of follow-up will be 15 years for each patient. At the end of the 15-year follow-up, the data will be stored for an additional 10 years before being deleted. Data will be recorded if the patients are willing to comply with the annual data collection. Should the DiMe Project be terminated at one stage, the data will be stored for 10 years after termination of the project before being deleted.

ELIGIBILITY:
Inclusion Criteria:

* symptomatic DM confirmed by a senior orthopedic surgeon based on physical examination and MRI
* age less than eighteen years
* informed consent freely granted and acquired before the start of the study from legal representative

Exclusion Criteria:

* concomitant or previous knee surgeries
* concomitant ligament knee injury that requires a surgical treatment
* concomitant fractures
* inflammatory or arthritic diseases.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children diagnosed with symptomatic DM confirmed on the basis of physical examination and MRI
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-09-08 (Actual); Primary Completion 2042-09-01 (Estimated); Study Completion 2042-09-01 (Estimated)

PRIMARY OUTCOMES:
Pedi-IKDC (0-100) among the three types of DM according to Ahn classification. | Enrollment period (approximately 5 years)

SECONDARY OUTCOMES:
Time to return to sport (months) among the three types of DM tear according to Ahn classification. | Entire study duration (approximately 20 years)
Tegner activity level scale (0-10) among the three types of DM tear according to Ahn classification. | Entire study duration (approximately 20 years)
  Tegner activity level scale:0=Sick leave or disability pension because of knee problems 10=Competitive sports Soccer - national and international elite

OTHER OUTCOMES:
Surgical treatment in each type of DM, according to Watanabe and Ahn classifications | Enrollment period (approximately 5 years)
Pedi-IKDC related to anthropometric features and anamnestic characteristics. | Enrollment period (approximately 5 years)
  The Pediatric International Knee Documentation Committee (Pedi-IKDC) Subjective Knee Evaluation Form
DM healing (timing of early phase, remodeling (high tissue enhancement), maturation measured in months from surgery - all measured with serial MRIs) | Entire study duration (approximately 20 years)

CONTACTS AND LOCATIONS:
Locations (12):
- Universitair Ziekenhuis, Leuven, Belgium
- Oulu University Hospital,, Oulu, Finland
- France (3):
  - CHU Grenoble, Grenoble
  - Clinique Rive Gauche, Toulouse
  - Department of Orthopaedic Surgery, Hôpital des Enfants, CHU de Toulouse, Toulouse
- Italy (2):
  - Policlinico San Pietro, Bergamo, BG
  - ASST Monza - Ospedale San Gerardo, Monza
- Portugal (2):
  - Department of Pediatric Orthopaedics, Hospital Pediátrico de -Coimbra, Coimbra
  - Hospital Cuf Descobertas, Lisbon
- Centre hospitalier universitaire vaudois (CHUV), Lausanne, Switzerland
- United Kingdom (2):
  - London Children's Hospital, London
  - SHEFFIELD CHILDREN'S NHS NHS Foundation Trust,, Sheffield

REFERENCES:
- [Background] Turati M, Anghilieri FM, Accadbled F, Piatti M, Di Benedetto P, Moltrasio F, Zatti G, Zanchi N, Bigoni M. Discoid meniscus in human fetuses: A systematic review. Knee. 2021 Jun;30:205-213. doi: 10.1016/j.knee.2021.04.006. Epub 2021 May 1. PMID 33945980
- [Background] Ahn JH, Lee SH, Yoo JC, Lee YS, Ha HC. Arthroscopic partial meniscectomy with repair of the peripheral tear for symptomatic discoid lateral meniscus in children: results of minimum 2 years of follow-up. Arthroscopy. 2008 Aug;24(8):888-98. doi: 10.1016/j.arthro.2008.03.002. Epub 2008 May 5. PMID 18657737
- [Background] Wasser L, Knorr J, Accadbled F, Abid A, Sales De Gauzy J. Arthroscopic treatment of discoid meniscus in children: clinical and MRI results. Orthop Traumatol Surg Res. 2011 May;97(3):297-303. doi: 10.1016/j.otsr.2010.11.009. Epub 2011 Mar 23. PMID 21435965
- [Background] Kinugasa K, Hamada M, Yonetani Y, Matsuo T, Mae T, Nakata K, Horibe S. Discoid lateral meniscal repair without saucerization for adolescents with peripheral longitudinal tear. Knee. 2019 Jun;26(3):803-808. doi: 10.1016/j.knee.2019.03.007. Epub 2019 May 7. PMID 31076246
- [Background] Matsuo T, Kinugasa K, Sakata K, Ohori T, Mae T, Hamada M. Post-operative deformation and extrusion of the discoid lateral meniscus following a partial meniscectomy with repair. Knee Surg Sports Traumatol Arthrosc. 2017 Feb;25(2):390-396. doi: 10.1007/s00167-016-4393-6. Epub 2016 Dec 23. PMID 28012004
- [Background] Nepple JJ, Milewski MD, Shea KG. Research in Osteochondritis Dissecans of the Knee: 2016 Update. J Knee Surg. 2016 Oct;29(7):533-538. doi: 10.1055/s-0036-1586723. Epub 2016 Aug 17. PMID 27532280
- [Background] Moksnes H, Engebretsen L, Seil R. The ESSKA paediatric anterior cruciate ligament monitoring initiative. Knee Surg Sports Traumatol Arthrosc. 2016 Mar;24(3):680-7. doi: 10.1007/s00167-015-3746-x. Epub 2015 Aug 7. PMID 26249112
- [Background] Scott EJ, Westermann R, Glass NA, Hettrich C, Wolf BR, Bollier MJ. Performance of the PROMIS in Patients After Anterior Cruciate Ligament Reconstruction. Orthop J Sports Med. 2018 May 25;6(5):2325967118774509. doi: 10.1177/2325967118774509. eCollection 2018 May. PMID 29854864
- [Background] Grant-Beuttler M, Jennings J, McCauley C, Dulay R, Grossnickle K, Kill K, Hay J. Development of an Electronic Version of The Children's Self-Perceptions of Adequacy in and Predilection for Physical Activity (CSAPPA) Scale. Pediatr Exerc Sci. 2017 Feb;29(1):153-160. doi: 10.1123/pes.2016-0115. Epub 2016 Oct 21. PMID 27768553
- [Background] Briggs KK, Lysholm J, Tegner Y, Rodkey WG, Kocher MS, Steadman JR. The reliability, validity, and responsiveness of the Lysholm score and Tegner activity scale for anterior cruciate ligament injuries of the knee: 25 years later. Am J Sports Med. 2009 May;37(5):890-7. doi: 10.1177/0363546508330143. Epub 2009 Mar 4. PMID 19261899
- [Background] Dietvorst M, Reijman M, van Groningen B, van der Steen MC, Janssen RPA. PROMs in paediatric knee ligament injury: use the Pedi-IKDC and avoid using adult PROMs. Knee Surg Sports Traumatol Arthrosc. 2019 Jun;27(6):1965-1973. doi: 10.1007/s00167-017-4687-3. Epub 2017 Sep 19. PMID 28929208
- [Background] Outerbridge RE. The etiology of chondromalacia patellae. 1961. Clin Orthop Relat Res. 2001 Aug;(389):5-8. doi: 10.1097/00003086-200108000-00002. No abstract available. PMID 11501822
- [Background] CholeS Study Group, West Midlands Research Collaborative. Population-based cohort study of outcomes following cholecystectomy for benign gallbladder diseases. Br J Surg. 2016 Nov;103(12):1704-1715. doi: 10.1002/bjs.10287. Epub 2016 Aug 26. PMID 27561954
- [Background] Courtney A, O'Connell R, Rattay T, Kim B, Cutress RI, Kirwan CC, Gandhi A, Fairbrother P, Sharma N, Cartlidge CWJ, Horgan K, McIntosh SA, Leff DR, Vidya R, Potter S, Holcombe C, Copson E, Coles CE, Dave RV. The B-MaP-C study: Breast cancer management pathways during the COVID-19 pandemic. Study protocol. Int J Surg Protoc. 2020;24:1-5. doi: 10.1016/j.isjp.2020.07.003. Epub 2020 Jul 29. PMID 32838092